CLINICAL TRIAL: NCT00545545
Title: A Phase 1b, Safety, PK, and Efficacy, Multicenter, Dose-Escalating Study of Imprime PGG in Combination With Cetuximab With and Without Irinotecan Therapy in Patients With Recurrent/Progressive Colorectal Carcinoma Following Treatment With a 5-FU Regimen.
Brief Title: Safety/Efficacy Study of Imprime PGG With Cetuximab in Patients With Recurrent/Progressive Colorectal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-CL-PGG-CRC0713
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Colorectal Carcinoma; Progressive Colorectal Carcinoma
Keywords: Colorectal; Carcinoma; Recurrent; Progressive; Cetuximab; Irinotecan; 5-Fluorouracil
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma; Recurrence | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Imprime PGG 2mg/kg+Cetuximab+Irinotecan (Experimental): Treatment Arm 1 2.0 mg/kg Imprime PGG administered weekly with combination therapy of cetuximab and irinotecan.
  Interventions: Biological: Imprime PGG 2 mg/kg; Biological: Cetuximab; Drug: Irinotecan
- Imprime PGG 4mg/kg+Cetuximab+Irinotecan (Experimental): Treatment Arm 1 4.0 mg/kg Imprime PGG administered weekly with combination therapy of cetuximab and irinotecan.
  Interventions: Biological: Imprime PGG 4 mg/kg; Biological: Cetuximab; Drug: Irinotecan
- Imprime PGG 6mg/kg+Cetuximab+Irinotecan (Experimental): Treatment Arm 1 6.0 mg/kg Imprime PGG administered weekly with combination therapy of cetuximab and irinotecan.
  Interventions: Biological: Cetuximab; Drug: Irinotecan; Biological: Imprime PGG 6mg/kg
- Imprime PGG 2mg/kg+Cetuximab (Experimental): Treatment Arm 2 2.0 mg/kg Imprime PGG administered weekly with concomitant cetuximab.
  Interventions: Biological: Imprime PGG 2 mg/kg; Biological: Cetuximab
- Imprime PGG 4mg/kg+Cetuximab (Experimental): Treatment Arm 2 4.0 mg/kg Imprime PGG administered weekly with concomitant cetuximab.
  Interventions: Biological: Imprime PGG 4 mg/kg; Biological: Cetuximab
- Imprime PGG 6mg/kg+Cetuximab (Experimental): Treatment Arm 2 6.0 mg/kg Imprime PGG administered weekly with concomitant cetuximab.
  Interventions: Biological: Cetuximab; Biological: Imprime PGG 6mg/kg

INTERVENTIONS:
Biological: Imprime PGG 2 mg/kg — Infusion of 2mg/kg on Day 1 of each week for 6 weeks (one cycle) Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Imprime PGG 2mg/kg+Cetuximab; Imprime PGG 2mg/kg+Cetuximab+Irinotecan
Biological: Imprime PGG 4 mg/kg — Infusion of 4mg/kg on Day 1 of each week for 6 weeks (one cycle). Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Imprime PGG 4mg/kg+Cetuximab; Imprime PGG 4mg/kg+Cetuximab+Irinotecan
Biological: Cetuximab — Infusion 400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
Drug: Irinotecan — Infusion 125 mg/m2 i.v. over 1.5 hours on Days 1, 8, 15, and 22 of each 6-week treatment cycle
  Arms: Imprime PGG 2mg/kg+Cetuximab+Irinotecan; Imprime PGG 4mg/kg+Cetuximab+Irinotecan; Imprime PGG 6mg/kg+Cetuximab+Irinotecan
Biological: Imprime PGG 6mg/kg — Infusion of 6mg/kg on Day 1 of each week for 6 weeks (one cycle) Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Imprime PGG 6mg/kg+Cetuximab; Imprime PGG 6mg/kg+Cetuximab+Irinotecan

SUMMARY:
Phase 1b, safety, pharmacokinetic, and efficacy, multicenter, dose-escalating Study of Imprime PGG™ Injection dosed in combination with Cetuximab and concomitant irinotecan therapy. Enrolled patients will have a confirmed diagnosis of recurrent or progressive colorectal carcinoma following treatment with a 5-fluorouracil-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Is between the ages of 18 and 75 years old, inclusive;
2. Has a recurrent or progressive carcinoma of the colon or rectum with documented histological confirmation of primary carcinoma;
3. Has measurable disease, defined as at least one tumor that fulfills the criteria for a target lesion according to RECIST;
4. Has previously received treatment with 5-FU, alone or in combination with other anti-tumor medications (except as in exclusion #1 below); Prior treatment with capecitabine (Xeloda®) will be considered to fulfill the requirement for prior treatment with 5-FU;
5. Has a Karnofsky Score of ≥ 70;
6. Has a life expectancy of > 3 months;
7. Has adequate bone marrow reserve as evidenced by:

   1. ANC ≥ 1,500/μL
   2. PLT ≥ 100,000/μL
   3. HGB ≥ 9 g/dl;
8. Has adequate renal function as evidenced by serum creatinine ≤ 1.5X the upper limit of normal (ULN) for the reference lab;
9. Has adequate hepatic function as evidenced by:

   1. Serum total bilirubin ≤ 1.0 mg/dL
   2. AST ≤ 3X ULN for the reference lab (≤ 5X ULN for patients with known hepatic metastases)
   3. ALT ≤ 3X ULN for the reference lab (≤ 5X ULN for patients with known hepatic metastases);
10. Has discontinued any CYP3A4 enzyme-inducing anticonvulsants (such as phenytoin, phenobarbital or carbamazepine) and antimicrobials (such as refampin and rifabutin), St. John's Wort, and ketoconasole at least two weeks prior to Day 1
11. Has recovered from the effects of any prior surgery, radiotherapy, or chemotherapy;
12. Has read, understood and signed the informed consent form (ICF) approved by the Independent Review Board/Ethics Committee (IRB/EC); and
13. If a woman of childbearing potential or a fertile man (and his partners), must agree to use an effective form of contraception during the study and for 120 days following the last dose of study medication (an effective form of contraception is an hormonal contraceptive or a double-barrier method).

Exclusion Criteria:

1. Has previously received treatment with cetuximab or irinotecan;
2. Has a known hypersensitivity to cetuximab, murine proteins, or any component of cetuximab;
3. Has a hereditary fructose intolerance;
4. Has a known hypersensitivity to baker's yeast, or has an active yeast infection;
5. Has had previous exposure to Betafectin® or Imprime PGG;
6. Has received previous radiation therapy to >30% of active bone marrow;
7. Has a fever of >38.5º C within 3 days prior to initial dosing;
8. Has known or suspected central nervous system (CNS) metastases;
9. Had a second malignancy within the previous 5 years, except for basal cell carcinoma, cervical intra-epithelial neoplasia or curatively-treated prostate cancer with a PSA of < 2.0 ng/mL;
10. Has known HIV/AIDS, Hepatitis B, Hepatitis C, connective tissue or autoimmune disease, or other clinical diagnosis, ongoing or intercurrent illness that in the investigator's opinion would prevent participation;
11. If female, is pregnant or breast-feeding;
12. Is receiving concurrent investigational therapy or has received investigational therapy within a period of 30 days prior to the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory-authority-approved indication); or
13. Has previously received an organ or progenitor/stem cell transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Belen Tamayo, MD, Principal Investigator — The Medical City Hospital; Gerardo Cornelio, MD, FPCP/FPS, Principal Investigator — Philippines General Hospital
Locations (2):
- Philippines (2):
  - Medical City, Makati City
  - Philippine General Hospital, Manila

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase 1b/2 dose-escalating (ascending dose model) design with 10 subjects enrolled in stage 1, 22 additional subjects in stage 2, for a total of 32 subjects enrolled sequentially into two treatment arms across Southeast Asia clinical sites.
  First subject enrolled: 15 Oct 2007 Last subject last visit: 04 Nov 2009
Pre-assignment Details: A total of 32 participants enrolled, all participants received at least one dose of study treatment.
Groups:
- Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan: Imprime PGG® infusion:
  2 mg/kg i.v. over 1 hr on Days 1, 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Cetuximab infusion:
  400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Irinotecan infusion:
  125 mg/m2 i.v. over 1.5 hours on Days 1, 8, 15, and 22 of each 6-week treatment cycle
- Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan: Imprime PGG® infusion:
  4 mg/kg i.v. over 2 hours on Days 1, 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Cetuximab infusion:
  400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Irinotecan infusion:
  125 mg/m2 i.v. over 1.5 hours on Days 1, 8, 15, and 22 of each 6-week treatment cycle
- Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan: Imprime PGG® infusion:
  6 mg/kg i.v. over 3 hours on Days 1, 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Cetuximab infusion:
  400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Irinotecan infusion:
  125 mg/m2 i.v. over 1.5 hours on Days 1, 8, 15, and 22 of each 6-week treatment cycle
- Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab: Imprime PGG® infusion:
  2 mg/kg i.v. over 1 hr on Days 1, 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Cetuximab infusion:
  400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle
- Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab: Imprime PGG® infusion:
  4 mg/kg i.v. over 2 hours on Days 1, 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Cetuximab infusion:
  400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle
- Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab: Imprime PGG® infusion:
  6 mg/kg i.v. over 3 hours on Days 1, 8, 15, 22, 29, and 36 of each 6-week treatment cycle;
  Cetuximab infusion:
  400 mg/m2 over 2 hours on Day 1, then 250 mg/m2 over 1 hour on Days 8, 15, 22, 29, and 36 of each 6-week treatment cycle
Period: Overall Study
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Started | 3 | 7 | 0 | 4 | 9 | 9
Discontinued | 3 | 7 | 0 | 4 | 9 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 0 | 4 | 9 | 9
Not completed — Progressive Neoplastic Disease | 1 | 5 | 0 | 4 | 8 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Irinotecan intolerance | 1 | 1 | 0 | 0 | 0 | 0
Not completed — No target lesions to track post surgery | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety population comprised all subjects who received any amount of Imprime PGG.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab | Total
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (6.6) | 52.9 (12.4) |  | 52.0 (10.8) | 52.6 (11.8) | 61.9 (9.3) | 55.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 1 | 4 | 2 | 10
  Male | 3 | 4 | 0 | 3 | 5 | 7 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  East Southeast Asian | 3 | 7 |  | 4 | 9 | 9 | 32
Baseline Karnofsky Performance Status Score [Mean (Standard Deviation); unit: units on a scale] — Karnofsky Performance Status Score:
  100-Normal no complaints; no evidence of disease 90-Carry on normal activity; minor signs of disease 80-Normal activity with effort; some signs of disease 70-Cares for self; unable to carry on normal activity or active work 60-Requires occasional assistance, can care for personal needs 50-Requires considerable assistance & frequent medical care 40-Disabled; requires assistance 30-Severely disabled; hospital admission indicated 20-Very sick; hospital admission & supportive treatment necessary 10-Moribund; fatal process progressing rapidly 0-Dead
  units on a scale | 86.7 (15.3) | 92.9 (7.6) |  | 92.5 (5.0) | 90.0 (7.1) | 93.3 (8.7) | 91.4 (8.6)
Baseline Height [Mean (Standard Deviation); unit: cm] | 168.3 (4.2) | 162.3 (11.6) |  | 163.3 (7.5) | 161.8 (9.0) | 162.1 (8.5) | 163.2 (9.1)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 69.5 (13.1) | 57.0 (15.1) |  | 60.2 (11.5) | 57.6 (11.6) | 63.4 (8.4) | 60.7 (12.7)
Baseline Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.8 (0.2) | 1.6 (0.3) |  | 1.6 (0.2) | 1.6 (0.2) | 1.7 (0.1) | 1.6 (0.3)
Time Since Initial Tumor Diagnosis [Mean (Standard Deviation); unit: days] | 630.7 (560.7) | 686.6 (354.7) |  | 710.5 (507.7) | 776.7 (597.1) | 526.6 (335.8) | 666.1 (436.1)
Initial Pathologic Diagnosis [Number; unit: participants]
  Colon Carcinoma | 2 | 2 |  | 2 | 5 | 8 | 19
  Rectum Carcinoma | 1 | 5 |  | 2 | 4 | 1 | 13
Basis of Diagnosis [Number; unit: participants]
  Cytology | 0 | 0 |  | 0 | 1 | 0 | 1
  Histology | 3 | 7 |  | 4 | 8 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Safety and Maximum Tolerated Dosage of Imprime PGG When Used in Combination With Cetuximab With or Without Irinotecan Therapy
Description: Safety and maximum tolerated dosage (MTD) of Imprime PGG was determined by the Adverse Events Task Force based on the drug-related adverse events experienced by subjects that met the criteria for a dose limiting toxicity (DLT) within a timeframe of the first 3 weeks of treatment and 1 week follow-up.
  If one in the initial three subjects for a dose group experienced a DLT, three additional subjects were enrolled in that dose group. If two or more subjects in the expanded dose group experienced a DLT, the study was to be stopped and the MTD was defined as the dose prior to the dose at which the DLT was observed. If a DLT occurred in the first dose group (2 mg/kg Imprime PGG), the protocol allowed for the next group to be dosed at a reduced dose of 1 mg/kg Imprime PGG.
  The dose groups described above were: Dose Group 1 (Imprime PGG 2 mg/kg), Dose Group 2 (Imprime PGG 4 mg/kg), Dose Group 3 (Imprime PGG 6 mg/kg).
Time Frame: From the date of the first dose of study drug to disease progression or until development of a drug toxicity that precludes further protocol treatment, up to 15 months
Population: The safety population comprised of all subjects who received any amount of Imprime PGG.
Measure: Number; unit: participants
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
participants
  Subjects Who Received Treatment | 3 | 7 |  | 4 | 9 | 9
  Subjects Who Discontinued the Study | 3 | 7 |  | 4 | 9 | 9

2. Secondary Outcome: Rate of Number of Participants With Tumor Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD) in Each Study Arm
Description: The best observed overall response rates were defined as the number of participants experiencing a best tumor response of either complete response (CR; disappearance of all target lesions), partial response (PR; >=30% decrease in the sum of diameters of target lesions), stable disease (SD) or progressive disease (PD) based on RECIST criteria v1.0.
Time Frame: From the date of the first dose of study drug to disease progression or last objective evaluation of the tumor before treatment discontinuation due to any reason, up to 15 months
Population: The ITT population is comprised of all subjects who have been enrolled in the study. All subjects were included in the Safety and ITT populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
Participants
  Number of participants with best response of CR | 0 | 0 |  | 0 | 0 | 0
  Number of participants with best response of PR | 2 | 1 |  | 0 | 3 | 2
  Number of participants with best response of SD | 1 | 6 |  | 3 | 3 | 2
  Number of participants with best response of PD | 0 | 0 |  | 1 | 3 | 4
  No information | 0 | 0 |  | 0 | 0 | 1

3. Secondary Outcome: Overall Response Rate (ORR) Per RECIST Criteria v1.0 in Each Study Arm
Description: The overall response rate was defined as the number of participants experiencing a best tumor response of either complete response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of diameters of target lesions) based on RECIST criteria v.1.0. Overall response rate (ORR) = CR + PR.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
Participants | 2 | 1 |  | 0 | 3 | 2

4. Secondary Outcome: Disease Control Rate (DCR) Per RECIST Criteria v1.0 in Each Study Arm
Description: The disease control rate was defined as the number of participants experiencing a best tumor response of either complete response (CR; disappearance of all target lesions), partial response (PR; >=30% decrease in the sum of diameters of target lesions) or stable disease (SD) based on RECIST criteria v.1.0. Disease control rate (DCR) = CR + PR + SD.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
Participants | 3 | 7 |  | 3 | 6 | 4

5. Secondary Outcome: Duration of Time-to-Progression (TTP) in Each Study Arm
Description: Time-to-progression (TTP) was defined as the time from the date of the first dose of study drug to the date of the first documented progression (date of the CT scan where progression was first observed; or where progression was first observed if clinical assessment). Subjects who did not progress were censored at the last objective evaluation (the date of the last CT scan; or last observed clinical assessment).
Time Frame: The time from the date of the first dose of study drug to the date of the first documented progression or last objective evaluation of the tumor before treatment discontinuation due to any reason, up to 15 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
days | 204.0 [166.0 to 204.0] | 148.0 [131.0 to 194.0] |  | 101.5 [19.0 to 212.0] | 163.0 [46.0 to 208.0] | 61.0 [38.0 to 250.0]

6. Secondary Outcome: Duration of Overall Tumor Response in Each Study Arm
Description: The duration of objective tumor response was defined as the time from the date of the first documented CT scan showing CR (disappearance of all target lesions) or PR (>=30% decrease in the sum of diameters of target lesions), whichever occurred first, to the date of the first documented progression (date of CT scan where PD was first observed; or where progression was first observed if based on a clinical assessment).
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
days | 149.5 [141.0 to 158.0] | 411.0 [141.0 to 411.0] |  | 0 [0.0 to 0.0] | 171.5 [169.0 to 174.0] | 99.0 [99.0 to 174.0]

7. Secondary Outcome: Duration of Disease Control in Each Study Arm
Description: Duration of stable disease (SD) was to be an efficacy variable, however, duration of disease control was used in place of duration of stable disease, as it is a more clinically meaning measure of the effectiveness of the treatment. Duration of disease control was defined as the time from the date of the first documented CT scan showing CR (disappearance of all target lesions), PR (>=30% decrease in the sum of diameters of target lesions) or SD, whichever occurred first, to the date of the first documented progression (date of CT scan where PD was first observed; or where progression was first observed if based on a clinical assessment).
Time Frame: The time from the date of first dose of study drug to the date of first documented progression, or last objective evaluation of the tumor before treatment discontinuation due to any reason, up to 15 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Number analyzed (Participants) | 3 | 7 | 0 | 4 | 9 | 9
days | 149.5 [141.0 to 158.0] | 93.5 [78.0 to 147.0] |  | 85.0 [39.0 to 172.0] | 148.0 [127.0 to 174.0] | 99.0 [43.0 to 211.0]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product to the discontinuation of study plus 30 days after the last dose of study drug or until the subject began alternative therapy, through end of treatment, up to 15 months
Description: The reason the number of participants at risk is zero for the 6 mg group in Arm 1 is that no patients were dosed in this group.
Arm/Group | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/7 | 0/0 | 2/4 | 4/9 | 2/9
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 0/0 | 4/4 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan (N=3) | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan (N=7) | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan (N=0) | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab (N=4) | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab (N=9) | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Perianal abscess (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Blood amylase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
International normalized ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Familial periodic paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Imprime PGG Injection 2 mg/kg+ Cetuximab + Irinotecan (N=3) | Arm 1, Imprime PGG Injection 4 mg/kg+ Cetuximab + Irinotecan (N=7) | Arm 1, Imprime PGG Injection 6 mg/kg+ Cetuximab + Irinotecan (N=0) | Arm 2, Imprime PGG Injection 2 mg/kg+ Cetuximab (N=4) | Arm 2, Imprime PGG Injection 4 mg/kg+ Cetuximab (N=9) | Arm 2, Imprime PGG Injection 6 mg/kg+ Cetuximab (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 2 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 3
Leukpoenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 6 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Otitis externa (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival cyst (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular surface disease (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 0 | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0
Perianal abscess (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Generalized muscle ache (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1 | 2 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 0 | 1 | 1
Viceral oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 0 | 3 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine amniotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Alanine amniotransferase increased (Investigations) | 1 | 4 | 0 | 3 | 5 | 3
Asparate amniotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Asparate amniotransferase increased (Investigations) | 0 | 4 | 0 | 2 | 6 | 4
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 3 | 3 | 3
Blood amylase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 3 | 5 | 0 | 3 | 2 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 1 | 3 | 4
Blood bicarbonate increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 3 | 0 | 3 | 3 | 4
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Blood magnesium increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 4 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Blood urea nitrogen/creatinine ratio decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 1 | 3 | 3
Creatine phosphokinase decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram poor r-wave progression (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gammaglutamyltransferase increased (Investigations) | 1 | 5 | 0 | 3 | 4 | 4
Globulins increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 2
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 6 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1 | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 5 | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6 | 0 | 1 | 7 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 2 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 4 | 0 | 1 | 3 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0
Nitrate urine present (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1
Genital haemorhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 0 | 0 | 0
Carbuncle (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatits acneform (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 3 | 8 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 6 | 2
Excoriation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythordysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Phelbitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less